CLINICAL TRIAL: NCT03217175
Title: Efficacy of Glucagon In the Prevention of Hypoglycemia During Mild Exercise
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of appropriate funds
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Steven J. Russell, MD, PhD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2017P001409
Record Dates: First submitted 2017-07-10; First posted 2017-07-13 (Actual); Results first posted 2019-11-18 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-11

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: bionic pancreas; type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Glucagon

STUDY DESIGN:
Intervention Model Description: Once the subject has been enrolled and eligibility of subjects has been established, subjects will be randomized to one of the possible two visit-orders. In random order, subjects will complete an insulin only exercise visit and a bi-hormonal exercise visit. The outpatient run-in period for both exercise visits will use the bi-hormonal bionic pancreas.
Who Masked: Participant
Masking Description: The study will be performed in single-blind fashion in that the participant will not know whether the bionic pancreas glucagon pump is filled with glucagon or placebo during the exercise visits. Study staff will fill the tandem t:slim glucagon pump with either glucagon or placebo according to the subject's randomization order. The subject will not be aware of their randomization. New infusion sets for both the glucagon/placebo and insulin pumps will be placed using an FDA approved steel cannula infusion set.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Bihormonal Bionic Pancreas (Active Comparator): Bihormonal bionic pancreas exercise visit - subjects will participate in the outpatient bihormonal bionic pancreas run in period, and will use the bihormonal bionic pancreas for their exercise visit at the end of the run in. The glucagon pump of the bionic pancreas will be filled with glucagon.
  Interventions: Device: Bihormonal Bionic Pancreas; Drug: Glucagon
- Insulin Only Bionic Pancreas (Placebo Comparator): Insulin-only bionic pancreas exercise visit - Bihormonal bionic pancreas exercise visit - subjects will participate in the outpatient bihormonal bionic pancreas run in period, and will use the insulin-only bionic pancreas for their exercise visit at the end of the run in. The glucagon pump of the bionic pancreas will be filled with placebo (normal saline).
  Interventions: Device: Insulin Only Bionic Pancreas; Drug: Placebo

INTERVENTIONS:
Device: Bihormonal Bionic Pancreas — The glucagon pump will be filled with glucagon during the exercise visit
  Arms: Bihormonal Bionic Pancreas
Device: Insulin Only Bionic Pancreas — The glucagon pump will be filled with placebo during the exercise visit, and the bionic pancreas will operate in an insulin only mode.
  Arms: Insulin Only Bionic Pancreas
Drug: Glucagon — Glucagon will be given according to the algorithm in the bihormonal bionic pancreas
  Arms: Bihormonal Bionic Pancreas
Drug: Placebo — Placebo will be given instead of glucagon according to the algorithm in the insulin-only bionic pancreas
  Arms: Insulin Only Bionic Pancreas

SUMMARY:
The study will consist of two study arms. Each arm will include a 24-96 hour outpatient run-in period prior to their exercise visit wearing the bi-hormonal bionic pancreas. In random order subjects will then complete two approximately 5-hour exercise visits, one wearing the bi-hormonal bionic pancreas and one wearing the insulin-only bionic pancreas.

DETAILED DESCRIPTION:
Twenty subjects will participate in two experimental periods. Each will include a 24-96 hour outpatient run-in period prior to their exercise visit wearing the bi-hormonal bionic pancreas. This will allow the bionic pancreas to adapt to their diabetes management needs. After the run-in period is complete, the subjects will participate in an exercise visit during which they will arrive fasting and remain fasted until the visit is completed. Subjects will walk on a treadmill for up to 1 hour at a comfortable walking pace. Plasma glucose (PG) measurements will be performed frequently. In one experimental period the bionic pancreas will remain in the bihormonal configuration and will deliver glucagon as needed during the exercise visit. In the other experimental period the glucagon will be replaced with a placebo during the exercise visit. The two experimental periods will be performed in random order. The study will be performed in single-blind fashion in that the participant will not know whether the bionic pancreas glucagon pump is filled with glucagon or placebo during the exercise visits. The outpatient run-in period will always be with the bi-hormonal bionic pancreas delivering glucagon.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and have had clinical type 1 diabetes for at least one year
* Diabetes managed using an insulin pump for ≥ 6 months
* Have used a CGM for ≥ 4 weeks over the last 12 months (usage does not need to be consecutive)
* Prescription medication regimen stable for > 1 month (except for medications that will not affect the safety of the study and are not expected to affect any outcome of the study, in the judgment of the principal investigator)
* Live within 120 minute radius of Massachusetts General Hospital
* Willing to remain within a 250 mile radius of the central monitoring location during the outpatient run-in period. No air travel will be allowed, and subjects will still be expected to follow the visit schedule as described.
* Willing to spend the night prior to both exercise visits in a hotel and fast overnight prior to exercise
* Willing to wear two steel cannula infusion sets (6 mm Contact Detach) and one Dexcom CGM sensor and change sets frequently (a new glucagon infusion set daily and a new insulin infusion set every other day during the outpatient run-in period)
* Have a mobile phone they will have access to at all times during the outpatient run-in period for making contact with study staff

Exclusion Criteria:

* Unable to provide informed consent (e.g. impaired cognition or judgment)
* Unable to safely comply with study procedures and reporting requirements (e.g. impairment of vision or dexterity that prevents safe operation of the bionic pancreas, impaired memory, unable to speak and read English)
* Current participation in another diabetes-related clinical trial that, in the judgment of the principal investigator, will compromise the results of this study or the safety of the subject
* Pregnancy (positive urine HCG), breast feeding, plan to become pregnant in the immediate future, or sexually active without use of contraception

  * Subjects must use acceptable contraception for the two weeks prior to the study, throughout the study and for the two weeks following the study.
  * Acceptable contraception methods include:Oral contraceptive pill (OCP), Intrauterine Device (IUD, hormonal or copper), Male condoms, Female condoms, Diaphragm or cervical cap with spermicide, Contraceptive patch (such as OrthoEvra), Contraceptive implant (such as Implanon, Nexplanon), Vaginal ring (such as NuvaRing), Progestin shot (such as Depo-Provera), Male partner with a vasectomy proven to be effective by semen analysis
* Current alcohol abuse (intake averaging > 3 drinks daily in last 30 days) or other substance abuse (use within the last 6 months of controlled substances other than marijuana without a prescription)
* Unwilling or unable or to avoid use of drugs that may dull the sensorium, reduce sensitivity to symptoms of hypoglycemia, or hinder decision making during the period of participation in the study (use of beta blockers will be allowed as long as the dose is stable and the subject does not meet the criteria for hypoglycemia unawareness while taking that stable dose, but use of benzodiazepines or narcotics or other central nervous system depressants, even if by prescription, may be excluded according to the judgment of the principal investigator)
* History of liver disease that is expected to interfere with the anti-hypoglycemia action of glucagon (e.g. liver failure or cirrhosis). Other liver disease (i.e. active hepatitis, steatosis, active biliary disease, any tumor of the liver, hemochromatosis, glycogen storage disease) may exclude the subject if it causes significant compromise to liver function or may do so in an unpredictable fashion.
* Renal failure requiring dialysis
* Personal history of cystic fibrosis, severe pancreatitis, pancreatic tumor, pancreatectomy or any other pancreatic disease leading to diabetes mellitus.
* Any known history of coronary artery disease including, but not limited to, history of myocardial infarction, stress test showing ischemia, history of angina, or history of intervention such as coronary artery bypass grafting, percutaneous coronary intervention, or enzymatic lysis of a presumed coronary occlusion)
* Abnormal EKG consistent with coronary artery disease or increased risk of malignant arrhythmia including, but not limited to, evidence of active ischemia, prior myocardial infarction, proximal LAD critical stenosis (Wellen's sign), prolonged QT interval (> 440 ms). Non-specific ST segment and T wave changes are not grounds for exclusion in the absence of symptoms or history of heart disease. A reassuring evaluation by a cardiologist after an abnormal EKG finding may allow participation.
* Congestive heart failure (established history of CHF, lower extremity edema, paroxysmal nocturnal dyspnea, or orthopnea)
* History of TIA or stroke
* Seizure disorder, history of any non-hypoglycemic seizure within the last two years, or ongoing treatment with anticonvulsants
* History of hypoglycemic seizures (grand-mal) or coma in the last year
* History of pheochromocytoma: fractionated metanephrines will be tested in patients with history increasing the risk for a catecholamine secreting tumor:

  * Episodic or treatment refractory (requiring 4 or more medications to achieve normotension) hypertension
  * Paroxysms of tachycardia, pallor, or headache
  * Personal or family history of MEN 2A, MEN 2B, neurofibromatosis, or von Hippel-Lindau disease
  * Adrenal tumor that has not undergone characterization for endocrine function
* Hypertension with systolic BP ≥160 mm Hg or diastolic BP ≥100 despite treatment
* Untreated or inadequately treated mental illness (indicators would include symptoms such as psychosis, hallucinations, mania, and any psychiatric hospitalization in the last year), or treatment with anti-psychotic medications that are known to affect glucose regulation.
* Electrically powered implants (e.g. cochlear implants, neurostimulators) that might be susceptible to RF interference
* Unable to completely avoid acetaminophen for duration of study
* History of adverse reaction to glucagon (including allergy) besides nausea and vomiting
* Established history of allergy or severe reaction to adhesive or tape that must be used in the study
* History of eating disorder within the last 2 years, such as anorexia, bulimia, or diabulemia or omission of insulin to manipulate weight
* History of intentional, inappropriate administration of insulin leading to severe hypoglycemia requiring treatment
* Use of oral (e.g. thiazolidinediones, biguanides, sulfonylureas, glitinides, DPP-4 inhibitors, SGLT-2 inhibitors) or non-insulin injectable (GLP-1 agonists, amylin) anti-diabetic medications
* Lives in or frequents areas with poor Verizon wireless network coverage (which would prevent remote monitoring)
* Hemoglobin < 12 g/dl for men, < 11 g/dl for women
* Any factors that, in the opinion of the principal investigator would interfere with the safe completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-08-18 (Actual); Primary Completion 2018-03-09 (Actual); Study Completion 2018-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Russell, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH Diabetes Research Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 22 subjects signed the consent form and screened into the study. 5 subjects were randomized and participated in the outpatient run-in period for one arm. Only 2 subjects of those 5 completed the arm. No subjects completed both arms of the study.
Groups:
- Bihormonal Bionic Pancreas First, Then Insulin-Only; Insulin Only Bionic Pancreas First, Then Bihormonal: Insulin-only bionic pancreas exercise visit - subjects will participate in the outpatient bionic pancreas run in period, and will use the insulin-only bionic pancreas for their exercise visit at the end of the run in. The glucagon pump of the bionic pancreas will be filled with placebo (normal saline).
  Placebo: Placebo will be given instead of glucagon according to the algorithm in the insulin-only bionic pancreas
  Bihormonal bionic pancreas exercise visit - subjects will participate in the outpatient bionic pancreas run in period, and will use the bihormonal bionic pancreas for their exercise visit at the end of the run in. The glucagon pump of the bionic pancreas will be filled with glucagon.
  Glucagon: Glucagon will be given according to the algorithm in the bihormonal bionic pancreas
Period: Overall Study
Arm/Group | Bihormonal Bionic Pancreas First, Then Insulin-Only | Insulin Only Bionic Pancreas First, Then Bihormonal
Started | 4 | 1
Completed | 0 | 0
Not Completed | 4 | 1
Not completed — Physician Decision | 4 | 1

BASELINE CHARACTERISTICS:
Population: All subjects enrolled in the study are included here. Most were not randomized prior to the study termination.
Groups:
- Whole Study: All subjects enrolled. The study was terminated before most subjects were able to be randomized.
Arm/Group | Whole Study
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.9 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22
Duration of diabetes [Mean (Standard Deviation); unit: years] | 21.4 (16.4)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Plasma Glucose < 60 mg/dl
Description: Number of subjects discordant between insulin-only and bihormonal bionic pancreas visits for reaching plasma glucose less than 60 mg/dl for greater than 2 consecutive measurements
Time Frame: 1 day (last day of each study arm - exercise visit)
Population: The study was terminated without performing any analysis of the data. The study was terminated because of a lack of appropriate funding.
Arm/Group | Bihormonal Bionic Pancreas | Insulin Only Bionic Pancreas
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Duration of Plasma Glucose < 60 mg/dl
Description: The amount of time the subject's plasma glucose is less than 60 mg/dl during the exercise visit
Time Frame: 1 day (last day of each study arm - exercise visit)
Population: as for outcome 1
Arm/Group | Bihormonal Bionic Pancreas | Insulin Only Bionic Pancreas
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Nadir Plasma Glucose
Description: The lowest plasma glucose experienced during the exercise visit
Time Frame: 1 day (last day of each study arm - exercise visit)
Population: as for outcome 1
Arm/Group | Bihormonal Bionic Pancreas | Insulin Only Bionic Pancreas
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Area Over the Curve and < 60 mg/dl
Description: The area over the plasma glucose curve but less than the 60 mg/dl threshold during exercise visit (a measure of hypoglycemic exposure)
Time Frame: 1 day (last day of each study arm - exercise visit)
Population: as for outcome 1
Arm/Group | Bihormonal Bionic Pancreas | Insulin Only Bionic Pancreas
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Time From Exercise Start to Plasma Glucose < 60 mg/dl
Description: The time from the start of exercise to the first plasma glucose measurement < 60 mg/dl that is reached
Time Frame: 1 day (last day of each study arm - exercise visit)
Population: as for outcome 1
Arm/Group | Bihormonal Bionic Pancreas | Insulin Only Bionic Pancreas
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Both study arms lasting up to 4 days each
Groups:
- Bihormonal Bionic Pancreas: Adverse events for participants in the bihormonal bionic pancreas arm are reported here.
- Insulin-only Bionic Pancreas: Adverse events for participants in the insulin-only bionic pancreas arm are reported here.
Arm/Group | Bihormonal Bionic Pancreas | Insulin-only Bionic Pancreas
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

LIMITATIONS AND CAVEATS:
The study was terminated early, and no data was analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT03217175/Prot_SAP_000.pdf